CLINICAL TRIAL: NCT03026855
Title: To Demonstrate the Safety and Efficacy of Autologous Platelet Rich Plasma (PRP) for the Treatment of Chronic Non-Healing Ulcers
Brief Title: Autologous Platelet Rich Plasma (PRP) for the Treatment of Chronic Non-Healing Ulcers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TotipotentRX Cell Therapy Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TPRX/PRP/NHU/141005
Record Dates: First submitted 2017-01-04; First posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Ulcer
Keywords: Autologous PRP; Non-healing ulcer; Point-of-care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous PRP Gel and PRP Injection (Experimental): Autologous PRP will be prepared using an advanced rapid point-of-care technology, the Res-Q™ 60 PRP system at the patient's bed side. The Activator solution for PRP gel will be prepared by combining human thrombin (500 IU/ml) with 1% Calcium Chloride.
  Interventions: Biological: Autologous PRP Gel and PRP Injection

INTERVENTIONS:
Biological: Autologous PRP Gel and PRP Injection — Autologous PRP prepared using the Res-Q™ 60 PRP system from patient's whole blood, will be injected subcutaneously around the periphery of the wound/ulcer.
  Based on the wound size and area, autologous platelet gel obtained by spraying simultaneously equal volumes of PRP and activator solution (thrombin with calcium chloride) will be applied topically over the ulcer or wound.
  Single dose of PRP injections and application of PRP gel will be administered, only on the day of treatment.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of autologous PRP injection in combination with topical application of PRP gel in treating chronic or non-healing ulcers on lower extremity using a rapid, intra-operative, point-of-care technology at the patient's bedside.

DETAILED DESCRIPTION:
Platelet Rich Plasma (PRP) therapy is an innovative treatment that uses body's own cells to relieve pain and promote accelerated healing of Non-healing Foot Ulcer /Wound. The body's response to any tissue injury is to deliver platelets, which play an instrumental role in the normal healing process by secreting growth factors and attracting stem cells-critical components of the healing cascade.

Any wound or ulcer on skin that has been present for 4-5 weeks duration, without healing is called a non-healing ulcer. Non-healing ulcers include venous, arterial, diabetic, pressure and traumatic ulcers. Cellular therapies using Autologous Platelet Rich Plasma provides new options for wound healing. The efficacy of the treatment has been proven in surgical applications, in the treatment of severe burns and in transplantation of cells and tissues.

Local application of a solution of plasma enriched in platelets derived from the patient's blood intends to trigger the healing process in non-responsive chronic wound, increase the wound repair rate and reduce pain. PRP is a good option for non-healing wounds because it utilizes the body's natural healing processes to jump-start wound healing. Plasma which contains very valuable growth factors is separated from other blood components utilizing a point of care technology based on density gradient centrifugation. The platelet rich plasma is harvested and then activated by a mixture of human thrombin and calcium chloride for initiating the healing cascade followed by PRP injection directly into the ulcer/wound periphery or spread over a wound in the form of a PRP gel.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female 18 to 85 years of age
* Chronic or Non-healing ulcer of any etiology (venous, pressure, arterial or diabetic foot ulcer) which is at least 4 weeks old
* Index foot ulcer located on the plantar, medial or lateral aspect of the foot (including all toe surfaces)
* Wound area (length x width) measurement must be between 0.5 cm^2 and 10 cm^2, inclusive
* If more than one non-healing ulcers is present, the largest wound will be selected
* Index ulcer must be clinically non-infected
* Full-thickness ulcer without exposure of bone, muscle, ligament or tendon
* Written informed consent must be obtained from either the patient or the patients legally acceptable representative prior to enrollment

Exclusion Criteria:

* Patients with known sensitivity to components of the PRP kit (calcium chloride, thrombin, acid citrate dextrose solution A (ACD-A))
* Smokers and individuals with systemic disease or history of anticoagulant, immuno-suppressive or antibiotic therapy in the last 3 months
* Platelet count < 105 x 10^3/ uL (according to CBC)
* Hemoglobin level < 10 g/dL (according to CBC)
* Wound is clinically infected
* Presence of platelet dysfunction syndrome or critical thrombocytopenia
* Bleeding disorders, collagen vascular disease or severe cardiovascular disorder
* Any malignancy other than non-melanoma skin cancer
* Patient is currently receiving or has received radiation or chemotherapy within 3 months prior to treatment
* If female, patient is pregnant, nursing or plans to become pregnant during the duration of the study
* Subject has inadequate venous access for blood draw required for PRP preparation
* Any chronic condition requiring the use of systemic corticosteroids 30 days prior to study entry and anytime during the course of the study
* Subject is on dialysis or has uncontrolled sugar levels

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-06; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of Wound/ Ulcers Healed | 24 weeks
  The number of wound/ ulcers healed will be assessed by visual inspection of reduction in wound size at 24 weeks post PRP therapy

SECONDARY OUTCOMES:
Time to Ulcer Healing | 24 weeks
  The average time taken for the ulcers to heal post PRP administration
Reduction in Pain using VAS pain score | 24 weeks
  Improvement in Pain and discomfort following PRP therapy
Changes in Quality of Life using the SF-36 Questionnaire | 24 weeks
  Improvement in Quality of Life of the patients following PRP therapy
Number of participants with treatment-related Adverse Events | 24 weeks
  Safety of the treatment will be assessed by measuring the number of treatment related adverse events and adverse reactions during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Suhail N Bukhari, MBBS, DNB, Principal Investigator — Fortis Escorts Heart Institute and Research Centre
Locations (1):
- Fortis Escorts Heart Institute and Research Centre, Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suthar M, Gupta S, Bukhari S, Ponemone V. Treatment of chronic non-healing ulcers using autologous platelet rich plasma: a case series. J Biomed Sci. 2017 Feb 27;24(1):16. doi: 10.1186/s12929-017-0324-1. PMID 28241824